CLINICAL TRIAL: NCT00983892
Title: Web-based Support for Caregivers of Veterans Undergoing Chemotherapy
Brief Title: Care Partners: Web-based Support for Caregivers of Veterans Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michigan State University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIR 08-309
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
Keywords: Cancer; caregiver; pain; symptom; information technology; palliative care
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CarePartners+ (Experimental): Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive the intervention (Intervention = access to a caregiver Web site that updates them on patient's symptoms and provides tailored problem solving advice).
  Interventions: Behavioral: Caregiver website
- CarePartners- (No Intervention): Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive nothing (i.e. no access to the caregiver website, or 'intervention').

INTERVENTIONS:
Behavioral: Caregiver website — Website receives patient symptom assessment data from IVR and provides caregivers with weekly updates on patient status, allowing caregivers to access tailored symptom management advice and formulate an action plan.
  Other Names: Care Partners
  Arms: CarePartners+

SUMMARY:
Given the growing strain on the Veterans Administration resulting from increasing caseloads of cancer patients, interventions are badly needed that assist patients in managing their illness, improve quality of life and avoid acute episodes that result in urgent care use and increased mortality. Previous studies have found that cancer patients undergoing chemotherapy can effectively manage their own symptoms when monitored using automated telephone calls. Such technology, however, may challenge the number of Veterans who lack social support and/or independence. The goal was to develop and test a technology that not only monitors patients automatically by telephone, but also gives them self management advice and engages a friend or family member to serve as a CarePartner willing to play a limited role in identifying patient symptoms and psychosocial needs to reinforce self management and provide social support. The investigators found that this technology indeed helped patients better control their symptoms, especially when a caregiver participated in the program along with them.

DETAILED DESCRIPTION:
Cancer is a prevalent problem that causes much suffering among Veterans and their families. Most interventions to improve symptom control require Veterans to engage in activities such as managing medications, altering diets, or accessing outside resources that may be beyond their reach due to limitations in physical and mental functioning. Friends and family inside and outside of the Veteran's household can help, but often lack the skills and resources they need to do so.

"Cancer CarePartners" was designed to address these needs by providing cancer-stricken Veterans and their informal caregivers with the information they need to make effective management decisions, decrease symptom burden, and improve outcomes. Cancer CarePartners is a Web-enabled program that alerts caregivers of patients' symptoms and provides them with a framework for identifying problems, receiving structured advice, formulating a 'task list,' and following up with their patients as they receive chemotherapy. Specifically, Cancer CarePartners includes weekly, automated telephonic symptom assessment (ATSA) with self-management (SM) support to the Veteran paired with Web-based alerts to the caregiver pointing them to a website where s/he can obtain customized advice. A randomized control trial was conducted to test the efficacy of this program in controlling symptoms as well as improving adherence to chemotherapy.

Objectives

1) To determine if Veterans undergoing chemotherapy who receive Cancer CarePartners report significant improvement in the summed severity of symptoms (the sum of 0-10 severity across 8 core symptoms) compared to Veterans receiving symptom monitoring and self-management advice; secondarily, to determine if they experience better adherence to chemotherapy and utilization. (2) To determine if caregivers participating in the intervention provide significantly more social support to patients than do controls; secondarily, to determine if they experience more caregiver burden and distress than do controls. (3) To determine whether impacts on patients are mediated by mastery. (4) To determine whether impacts on caregivers are mediated by mastery.

Methods Consenting Veterans with solid tumors undergoing chemotherapy at one of three VAMCs (Ann Arbor, Loma Linda and Fargo) who reported at least one core symptom at a moderate level or higher and had a caregiver willing to enroll in the study were randomly assigned to either 10 weeks of Cancer CarePartners or 10 weeks of automated, telephonic symptom assessment (ATSA) with self management support. Arms were balanced for non-small cell lung cancer status and caregiver type. Patients and caregivers were surveyed at intake, 10, and 14 weeks. In addition, the investigators tracked patient participation with ATSA and (in the experimental arm) caregiver use of the Cancer CarePartners Website. The investigators reviewed all medical records for content of care received during the 14 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older, cognitively intact, English-speaking, able to hear, and own a telephone.
* Patients can have any solid tumor.
* Patients must be initiating IV cytotoxic chemotherapy and, if recurrent, have experienced a 1 month treatment free interval.
* Caregivers must be 18 years or older, cognitively intact, English-speaking, and able to hear/speak for interviews.
* Caregivers must have access to a telephone and computer with high speed internet access.

Exclusion Criteria:

* Patients will be excluded if they have a hematologic malignancy or are receiving bone marrow transplantation.
* Patients and caregivers will be excluded if they have an untreated serious mental illness or cognitive impairment, are institutionalized or enrolled in hospice (prior to trial), or plan on not receiving all care from VA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-10; Primary Completion 2014-04 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria J. Silveira, MD MA MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silveira MJ, Given CW, Cease KB, Sikorskii A, Given B, Northouse LL, Piette JD. Cancer Carepartners: Improving patients' symptom management by engaging informal caregivers. BMC Palliat Care. 2011 Nov 25;10:21. doi: 10.1186/1472-684X-10-21. PMID 22117890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a five year study from October 1 2009 to Sept 30 2014. Patients were recruited from three VA oncology practices: Ann Arbor, Fargo, and Loma Linda.
Groups:
- CarePartners +: Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive access to a Web site that updates them on patient's symptoms and provides tailored problem solving advice.
  Caregiver website: Website receives patient symptom assessment data from IVR and provides caregivers with weekly updates on patient status, allowing caregivers to access tailored symptom management advice and formulate an action plan.
- CarePartners -: Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive nothing.
Period: Overall Study
Arm/Group | CarePartners + | CarePartners -
Started | 66 | 68
Completed | 56 | 56
Not Completed | 10 | 12
Not completed — Withdrawal by Subject | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CarePartners + | CarePartners - | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Full Range); unit: years] | 64 [46 to 87] | 62 [29 to 82] | 63 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 57 | 63 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 55 | 55 | 110
  Unknown or Not Reported | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 42 | 48 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 15 | 33
Summed symptom severity [Mean (Standard Deviation); unit: units on a scale 0-80] — symptom severity = the sum across 8 core symptoms rated by the patient on a scale of 0 to 10 (higher is worse).
  units on a scale 0-80 | 27.8 (13.7) | 28.1 (16.6) | 28.0 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Summed Symptom Severity
Description: Summed severity across 8 symptoms of interest, as measured using the MD Anderson Symptom Inventory. 8 core symptoms rated by the patient on a scale of 0 to 10. These 8 symptoms were chosen based on their prevalence of 50% or greater in the population of interest. Higher scores mean WORSE or GREATER SYMPTOM BURDEN.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CarePartners Intervention +: Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive access to a Web site that updates them on patient's symptoms and provides tailored problem solving advice.
  Caregiver website: Website receives patient symptom assessment data from IVR and provides caregivers with weekly updates on patient status, allowing caregivers to access tailored symptom management advice and formulate an action plan.
- Control: Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive nothing.
Arm/Group | CarePartners Intervention + | Control
Number analyzed (Participants) | 66 | 68
units on a scale | 23.2 (16.4) | 19.9 (14.9)
Statistical Analysis 1: Comparison: CarePartners Intervention + vs Control; Test type: Superiority or Other; p = 0.030, GEE; Adjusting for baseline symptom severity, caregiver type, week number, and cancer site; Slope = -1.56, 95% CI 2-sided [-2.97 to -0.15]

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- CarePartners+: Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive access to a Web site that updates them on patient's symptoms and provides tailored problem solving advice.
  Caregiver website: Website receives patient symptom assessment data from IVR and provides caregivers with weekly updates on patient status, allowing caregivers to access tailored symptom management advice and formulate an action plan.
- CarePartners-: Patients receive automated telephonic symptom assessment and symptom management advice; caregivers receive nothing.
Arm/Group | CarePartners+ | CarePartners-
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68

LIMITATIONS AND CAVEATS:
Recruitment rates were lower than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes